CLINICAL TRIAL: NCT04473677
Title: A New Quantitative Fecal Immunochemical Test Can Improve Diagnostic Accuracy in Detecting Colorectal Advanced Adenoma.
Brief Title: A New Quantitative Fecal Immunochemical Test in Detecting Colorectal Advanced Adenoma
Status: Completed | Type: Observational
Sponsor: Shandong University (Other)
Responsible Party: Principal Investigator, Yanqing Li, Clinical Professor, Shandong University
Other Study IDs: 2020SDU-QILU-708
Record Dates: First submitted 2020-07-14; First posted 2020-07-16 (Actual); Last update posted 2021-06-18 (Actual); Status verified 2021-06

CONDITIONS: Colorectal Adenoma; Colorectal Neoplasm; Colorectal Cancer
Keywords: Colorectal Adenoma; Colorectal Neoplasms; Occult Bleeding; quantitative fecal immunochemical test; Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Colonoscopy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — stool samples
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Fecal Occult Blood Test: People in this group will detect hemoglobin in stool before colonoscopy by the new qFIT.
  Interventions: Diagnostic Test: The new qFIT and colonoscopy with pathological examination

INTERVENTIONS:
Diagnostic Test: The new qFIT and colonoscopy with pathological examination — Detect hemoglobin in stool by the new qFIT before colonoscopy, detect colon lesion using colonoscopy and pathological examination.

SUMMARY:
Early detecting and removing of colorectal advanced adenomas can reduce incidence of colorectal cancer. Because of the less bleeding of advanced adenomas, the sensitivity of existing quantitative fecal immunochemical test (qFIT) is unsatisfying. A new technology qFIT, which have a higher sensitivity in extremely low concentration of hemoglobin compared with existing commercially available qFIT, is developed and this study will prove the high diagnostic accuracy in detecting colorectal advanced adenoma.

DETAILED DESCRIPTION:
Colorectal cancer accounts for approximately 10% of all annually diagnosed cancers and cancer-related deaths worldwide. With progress of developing countries, it is predicted that the incidence of colorectal cancer worldwide will increase to 2.5 million new cases in 2035. The majority of colorectal cancer is thought to arise from precancerous lesions through the adenoma-carcinoma pathway. Detecting and removing of colorectal advanced adenomas can reduce incidence of colorectal cancer. Although colonoscopy is currently considered the most effective method for detecting advanced adenomas, individuals may be reluctant to undergo colonoscopy due to the uncomfortable feeling and the relatively high cost of colonoscopy. Conversely, stool tests are relatively cheap and more readily accepted. Annual fecal immunochemical test (FIT), one of the preferred methods of colorectal cancer screening, is economic and easy to use. However, the existing commercially available qFIT is insufficiently sensitive to the minor hemorrhage of advanced adenomas, and the sensitivity is about only 27% to 47%. To improve diagnostic accuracy in detecting colorectal advanced adenoma, an improved technology of qFIT, which have a higher sensitivity in extremely low concentration of hemoglobin in stool compared with existing commercially available qFIT, is developed. The investigators design this research to prove the diagnostic accuracy of the new qFIT in detecting colorectal advanced adenoma.

ELIGIBILITY:
Inclusion Criteria:

* 50-75 years old people;
* People sign an "informed consent form"

Exclusion Criteria:

* People with history of surgery in any part of the large bowel;
* People with history of colorectal cancer;
* People with history of other diseases that may produce fecal blood, such as active diverticulitis, inflammatory bowel disease, ischemic enteritis, vascular malformation of intestine, intestinal tuberculosis or Non-Hodgkin's lymphoma involving digestive tract;
* People with symptoms including visible rectal bleeding, hematuria, hemorrhoid bleeds, severe and acute diarrhea and 7th type stool (Bristol feces score);
* People are in pregnancy, lactation or menstrual phase;
* People with severe congestive heart failure or other sever disease cause cannot tolerate colonoscopy.

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Continuous participants intending to undergo colonoscopy and meet the inclusion and exclusion criteria from Qilu Hospital were enrolled.
Sampling Method: Probability Sample
Enrollment: 1600 (Actual)
Dates: Start 2020-08-17 (Actual); Primary Completion 2021-06-11 (Actual); Study Completion 2021-06-11 (Actual)

PRIMARY OUTCOMES:
The accuracy of the new qFIT to diagnose colorectal advanced adenoma. | 18 months
  The sensitivity, specificity, positive predictive value and negative predictive value.

SECONDARY OUTCOMES:
The accuracy of the new qFIT to diagnose colorectal cancer. | 18 months
  The sensitivity, specificity, positive predictive value and negative predictive value.
Develop a predictive model of advanced colorectal neoplasms which includes the value of qFIT. | 18 months
  Develop a predictive model of advanced colorectal neoplasms which includes the value of qFIT, age , sex, colorectal cancer family history, diet and so on.

CONTACTS AND LOCATIONS:
Overall Officials: Yanqing Li, PhD, Study Chair — Qilu Hospital of Shandong University
Locations (1):
- Qilu Hospital, Jinan, Shandong, China